CLINICAL TRIAL: NCT01769677
Title: A Randomized, Open-Label, 2-Period, Crossover Study to Assess the Bioequivalence of Two 45-mg and One 90-mg Hydrocodone Bitartrate Extended-Release Tablet
Brief Title: A Crossover Study to Assess the Bioequivalence of Hydrocodone Bitartrate Extended-Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C33237/1099
Record Dates: First submitted 2013-01-10; First posted 2013-01-17 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: Bioequivalence; Hydrocodone bitartrate extended-release tablets
MeSH Terms: conditions — Pain | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group AB (Experimental): Subjects in this group will receive study drug in the following sequence:
  * Treatment A: two 45-mg hydrocodone bitartrate extended-release tablets (reference).
  * Treatment B: one 90-mg hydrocodone bitartrate extended-release tablet (test).
  Interventions: Drug: 90 mg dose of the hydrocodone bitartrate extended-release tablet administered as either two 45-mg tablets (Treatment A) or one 90-mg tablet (Treatment B).
- Treatment Group BA (Experimental): Subjects in this group will receive study drug in the following sequence:
  * Treatment B: one 90-mg hydrocodone bitartrate extended-release tablet (test).
  * Treatment A: two 45-mg hydrocodone bitartrate extended-release tablets (reference).
  Interventions: Drug: 90 mg dose of the hydrocodone bitartrate extended-release tablet administered as either two 45-mg tablets (Treatment A) or one 90-mg tablet (Treatment B).

INTERVENTIONS:
Drug: 90 mg dose of the hydrocodone bitartrate extended-release tablet administered as either two 45-mg tablets (Treatment A) or one 90-mg tablet (Treatment B). — Each subject will receive 1 treatment during each administration period. Subjects will receive each of the 2 treatments once. There will be a minimum 14-day washout period between the 2 administrations of study drug. Treatments will be orally administered to subjects, while they are seated, at approximately 0800 (±2 hours) on the 1st day of each administration period.

SUMMARY:
The primary objective of this study is to assess the bioequivalence of two 45-mg hydrocodone bitartrate extended-release tablets and one 90-mg hydrocodone bitartrate extended-release tablet.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The subject can read, speak, and write in English.
* The subject is a man or woman 18 through 45 years of age, with a body mass index (BMI) of 20.0 to 30.0 kg/m2, inclusive.
* The subject is in good health as determined by medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
* Women must be surgically sterile, 2 years postmenopausal, or, if of child-bearing potential, be using an acceptable method of contraception, and agree to continued use of this method for the duration of the study and for 30 days after discontinuation of study drug. Acceptable methods of contraception include abstinence or an intrauterine device (known to have a failure rate of less than 1% per year).
* The subject has a negative alcohol test and urine drug screen.
* The subject must be willing and able to comply with study restrictions and to remain at the study center for the required duration of each study drug period during the study.

Exclusion Criteria:

* The subject has any clinically significant uncontrolled medical conditions (treated or untreated).
* The subject has a clinically significant deviation from normal in ECG or physical examination findings, as determined by the investigator or the medical monitor.
* The subject has habitually consumed, within the past 2 years, more than 21 units of alcohol per week, or has a history of alcohol, narcotic, or any other substance abuse as defined by the Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition, Text Revision (DSM-IV-TR, American Psychiatric Association 2000). NOTE: A unit of alcohol is equal to 1 ounce of hard liquor, 5 ounces of wine, or 8 ounces of beer.
* The subject is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including GI surgery; a history of appendectomy is allowed).
* The subject has received any investigational drug within 30 days or 5 half-lives (whichever is longer) before the 1st dose of study drug, or in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before the 1st dose of study drug.
* The subject has a known sensitivity or idiosyncratic reaction to hydrocodone or hydromorphone, their related compounds, or to any metabolites, or naltrexone, or any compound listed as being present in a study formulation.
* Other exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | Up to 72 hrs after each dose of study drug
  To assess the bioequivalence between 45-mg tablets and one 90-mg tablet of the hydrocodone bitartrate extended-release tablet.
Area under the plasma drug concentration by time curve AUC0-∞ | Up to 72 hrs after each dose of study drug
  To assess bioequivalence between two 45-mg tablets and one 90-mg tablet of the hydrocodone bitartrate extended-release tablet.

SECONDARY OUTCOMES:
Time to maximum observed plasma drug concentration (tmax) | Up to 72 hrs after each dose of study drug
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.
AUC from time 0 to 72 hours after study drug administration (AUC0-72) | Up to 72 hrs after each dose of study drug
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.
AUC from time 0 to the time of the last measurable drug concentration (AUC0-t) | Up to 72 hrs after each dose of study drug
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.
Percentage extrapolation, 100x(AUC0-∞-AUC0-t)/AUC0-∞) | Up to 72 hrs after each dose of study drug
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.
Apparent plasma terminal elimination rate constant (λz) and associated elimination half life (t½) | Up to 72 hrs after each dose of study drug
  To characterize the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.
Recording of Adverse Events | Adverse events will be collected for the duration of the study which is approximately 7 weeks
  To characterize the safety of the hydrocodone bitartrate extended-release tablet in healthy naltrexone-blocked subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 10470, Austin, Texas, United States